CLINICAL TRIAL: NCT06230783
Title: Connected Language and Speech Along the Spectrum of ADRD: Digital Assessment and Monitoring
Brief Title: Speech Pattern Evaluation and Analysis for Knowledge of AD
Acronym: SPEAK-AD
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Arizona State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2023-1740; 1R01AG082052-01 (NIH); A534255 (Other: UW Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW Madison); Protocol Version 10/14/2024 (Other: UW Madison)
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Wisconsin Alzheimer's Disease Research Center; Wisconsin Registry for Alzheimer's Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: TalkTracker — Participants will be asked to complete the speech collection procedures remotely/at home once per week for 8 weeks. The 8-week period of weekly remote speech collection will take place yearly for a total of 3 years. At the end of each 8-week study period for years 1-3, participants will complete a survey that asks questions about how easy/difficult the application was to use, how frustrated they felt using the application, and other usability questions.

SUMMARY:
The goal of this observational study is to validate changes in speech as a measure of cognition in individuals at increased risk of Alzheimer's disease and related dementias (ADRD). This study aims to clarify how speech may be affected by Alzheimer's disease.

Participants will complete speech collection sessions and a survey at home using an iPad. Participants can expect to be in the study for 3 years.

DETAILED DESCRIPTION:
Digital technology, including recorded speech, has the capability of providing a wealth of information about early changes to cognition and communication associated with developing Alzheimer's disease pathology, with the potential for highly accessible, yet low-burden measurement. In this project, researchers will recruit a subset of participants from two longitudinal, observational cohort studies enriched for individuals at risk for or living with Alzheimer's disease to record their speech at home with a mobile device, longitudinally. Our interdisciplinary team will then validate digital markers across all stages of Alzheimer's Disease and Related Dementias (ADRD), including the prodromal phase, and can enhance sensitivity and specificity of speech metrics while contributing valuable information about remote, noninvasive, and accessible assessment and disease monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in the Wisconsin Alzheimer's Disease Research Center (W-ADRC) Clinical Core or IMPACT studies, or in the Wisconsin Registry for Alzheimer's Prevention (WRAP)
* Cognitively unimpaired or have a diagnosis of Mild Cognitive Impairment (MCI)
* Ages 40-80 years
* Completion of a W-ADRC or WRAP study visit within the past or upcoming 12 months
* Have provided W-ADRC or WRAP with blood plasma Alzheimer's Disease

Exclusion Criteria:

* Not actively enrolled in W-ADRC or WRAP
* Diagnosis of dementia
* Impaired capacity or unwilling to consent
* Major neurological conditions
* Speech disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from the WRAP and W-ADRC studies
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Usability of remote at-home speech collection - objective | 3 years
  Usability will be measured objectively through the TalkTracker mobile application by obtaining compliance metrics (number of tasks completed, total number of errors, number of help requests).
Usability of remote at-home speech collection - objective | 3 years
  Usability will be measured objectively through the TalkTracker mobile application by obtaining compliance metric of time to completion.
Feasibility of remote at-home speech collection | 3 years
  Feasibility will be measured through numbers of retention, adherence, and accrual.
Feasibility of remote at-home speech collection | 3 years
  Feasibility will be measured through sample characteristics, and identification of productive recruitment methods.
Feasibility of remote at-home speech collection | 3 years
  Feasibility will be measured through identification of productive recruitment methods.
Usability of remote at-home speech collection - subjective | 3 years
  Subjective measurement usability will be assessed through the System Usability Scale (SUS) given to participants after each 8-week completion period. The SUS is a 7 item questionnaire, with a range of 1 to 5 (1 = strongly disagree, 5 = strongly agree). Higher scores on questions 1, 3, 5 and 7 indicate lower usability. Higher scores on questions 2, 4 and 6 indicate higher usability.

SECONDARY OUTCOMES:
Correlation between in-clinic speech metrics and remote at-home speech metrics | 3 years
  Correlation between in-clinic versus at-home speech samples will be measured by calculating the inter-class correlation and standard error of measurement on speech measures of interest (content information units, semantic relevance, words per minute). Determination of variance between in-person and at-home speech samples will be evaluated by analysis of covariance accounting for age, sex, education, and cognitive status.
Correlations between metrics from remote at-home speech and plasma amyloid-beta (pTau-217) | 3 years
  Correlations will be determined using mixed effects models examining change in speech measures over time with plasma amyloid-beta, covarying for age, sex and genetic risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly D Mueller, PhD, CCC-SLP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No